CLINICAL TRIAL: NCT02863250
Title: Improving Outcomes for Patients With Critical Bleeding Requiring Massive Transfusion
Brief Title: Australian and New Zealand Massive Transfusion Registry
Acronym: ANZ-MTR
Status: Recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: CSL Behring (Industry); Department of Health and Human Services Victoria (Unknown); National Blood Authority (Other); New Zealand Blood Service (Other)
Responsible Party: Principal Investigator, Erica Wood, Professor, Monash University
Other Study IDs: APP1074654
Record Dates: First submitted 2016-07-27; First posted 2016-08-11 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Massive Transfusion; Trauma; Cardiothoracic Surgery; Gastrointestinal Bleeding; Vascular Surgery; Obstetric Bleeding; Liver Transplant
MeSH Terms: conditions — Wounds and Injuries; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Massively transfused patients: Patients (18+ years) who have had a critical bleeding event that necessitated a massive transfusion (defined as 5 or more units of red cells in any 4 hour period)

SUMMARY:
Severe and un-stopped blood loss can occur for a number of different reasons including after a serious injury, delivery of a baby and following other medical and surgical emergencies. The investigators understanding of how to best treat people with serious bleeding is still incomplete, with many questions remaining. These include questions regarding how many people have serious bleeding events, what happens to them and the best way to treat them.

The Massive Transfusion Registry (MTR) is a register of patients who have experienced major blood loss that required a massive transfusion in any clinical setting.

The MTR uses electronic data extraction and data linkage methodologies. Pre-existing clinical data from hospital data sources, including Laboratory Information Systems (for transfusion history and laboratory results) and Health Information Services databases (for Patient demographics and admission data), are electronically extracted by staff employed at the participating hospitals. The data is then sent to the MTR Research Team, located at Monash University, where it is then linked, analysed and stored.

The establishment of a Massive Transfusion Registry will be a unique and important resource for clinicians in Australia, New Zealand and internationally, for Blood Services and for the broader community. It will provide valuable observational data regarding the types and frequency of conditions associated with critical bleeding requiring massive transfusion, the use of blood component therapy (i.e. ratios and quantities of different types of red cell to non- red cell components) and patient outcomes.

DETAILED DESCRIPTION:
The Australian and New Zealand Massive Transfusion Registry (ANZ-MTR) Clinical Dataset brings together data from multiple sources and analyses and reports contemporary information on transfusion practice and patient outcomes following critical bleeding (CB) and massive transfusion (MT) in all clinical settings, including surgery, trauma, obstetrics and gastrointestinal bleeding. Data on more than 6,000 patients from 25 participating sites have already been collected, analysed and results shared with participants.

The ANZ-MTR is a unique resource. Recognising the valuable dataset available for transfusion policy and practice improvement, the ANZ-MTR is now transitioning from primarily a research tool to a sustainable operational model to align with Australia's national safety and quality framework, whilst still allowing research opportunities.

ANZ-MTR data are already linked with the Australian and New Zealand National Death Indexes and the ANZ-MTR team is engaged with establishing linkages with other registries (e.g. intensive care, cardiothoracic surgery, trauma, maternity outcomes and others). This will provide expanded data for more sensitive outcome measurement.

The ANZ-MTR uses electronic data extraction and data linkage methodologies. Clinical data from hospital data sources, including Laboratory Information Systems (for transfusion history and laboratory results) and Health Information Services databases (for patient demographics and admission data), are electronically extracted by the participating hospitals. The data are then sent to the ANZ-MTR, located at Monash University, where the data from the separate information systems are linked to enable detailed analyses that otherwise would not be easily possible. Monash University's Department of Epidemiology and Preventive Medicine, where the ANZ-MTR is located, has internationally recognised expertise in the management and statistical analyses of large, complex electronic datasets.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over
* 5 or more units of red blood cells in any 4 hour period

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to participating hospitals, aged 18 years or over, who have had a critical bleeding event that necessitated a massive transfusion (defined as 5 or more units of red blood cells in any 4 hour period), in any clinical context.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2011-03; Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days

OTHER OUTCOMES:
Blood product use | 48 hours
  Trends in blood products transfused at 48 hours across various bleeding types

CONTACTS AND LOCATIONS:
Overall Officials: Erica Wood, MBBS, Principal Investigator — Monash University
Locations (1):
- Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No